CLINICAL TRIAL: NCT06000007
Title: Development and Implementation of a Behavioral Digital Therapeutic Designed to Support, Educate, Screen and Remotely Monitor Patients with Chronic Pain
Brief Title: Digital Therapeutic for Chronic Pain Feasibility Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Kari Stephens, Professor of Family Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00016340; 1R44AT011593-01 (NIH)
Record Dates: First submitted 2023-08-10; First posted 2023-08-21 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain
Keywords: chronic pain; primary care; digital therapeutic; mobile app; pain function; pain interference; psychotherapy
MeSH Terms: conditions — Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized control feasibility study with two arms: intervention arm vs. control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment as usual (Active Comparator): Treatment as usual arm entails the patients continuing to receive care from their primary care provider and any specialists they choose to get involved in their care.
  Interventions: Other: Treatment as usual
- Intervention arm (Active Comparator): Intervention arm includes access to the digital therapeutic mobile app in addition to treatment as usual
  Interventions: Device: 2Morrow Chronic Pain Self-Management Program - digital therapeutic mobile app

INTERVENTIONS:
Device: 2Morrow Chronic Pain Self-Management Program - digital therapeutic mobile app — 2Morrow Chronic Pain Self-Management Program is delivered via a mobile app that engaged patients in evidenced based psychotherapy for chronic pain, including Acceptance and Commitment Therapy and Cognitive Behavioral Therapy based activities, to improve a patient's pain self management. The mobile app also offers the ability to track activities, screen for other problems, support for communicating with medical providers, and access a coach via texting.
  Arms: Intervention arm
Other: Treatment as usual — Treatment as usual entails continuing with treatment for chronic pain with the patient's primary care provider and any potential specialists they choose to engage with.
  Arms: Treatment as usual

SUMMARY:
The investigators will conduct a 2-arm randomized control feasibility study to evaluate: 1) the feasibility of using the mobile app and an optional activity tracker, 2) the feasibility of conducting a 2-arm trial, and 3) estimate the effect size for planning for a larger efficacy trial based on our primary outcomes. The intervention arm will test a mobile app that aims to help people reduce pain interference who have chronic pain, as well as mental health issues with depression and anxiety. Participants in the intervention arm will also have the option to sense health data with a tracker that integrates with the app, which will inform the feasibility of this feature.

DETAILED DESCRIPTION:
This study will evaluate the existing 2Morrow Chronic Pain Self-Management Program, in the form of a mobile app, as a digital therapeutic for improving patients' pain self management and function who suffer from chronic pain. Specifically, the investigators will conduct a 2-arm randomized control feasibility study to evaluate: 1) the feasibility of using the mobile app and an optional activity tracker, 2) the feasibility of conducting a 2-arm trial, and 3) estimate the effect size for planning for a larger efficacy trial based on our primary outcomes. The intervention arm will test a mobile app that aims to help people reduce pain interference who have chronic pain, as well as mental health issues with depression and anxiety. Participants in the intervention arm will also have the option to sense health data with a tracker that integrates with the app, which will inform the feasibility of this feature.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years old
* at least one ICD pain related diagnosis noted in the electronic health record (EHR)
* at least 2 visits in a primary care clinic with at least one in the last 12 months
* willing to use a mobile app in English
* T-score for the PROMIS brief pain inventory of >= 55
* access to a smartphone
* willing to download and use a mobile app daily

Exclusion Criteria:

* current cancer related diagnosis (to exclude cancer related chronic pain)
* plans for surgery in next 3 months
* pregnant
* currently receiving hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
PROMIS Pain Interference Scale - Short Form 6b | will be measured at baseline, 1 month, 3 months, and 6 months after enrollment (and start of intervention in the intervention arm)
  Brief survey of patient's perceived pain interference in their ability to function; scores are normed on a T-score with 50 as the mean, 10 as the standard deviation, and higher scores are worse

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | will be measured at baseline, 1 month, 3 months, and 6 months after enrollment (and start of intervention in the intervention arm)
  depression symptom measure; scores range from 0 to 27; higher scores are worse
Generalized Anxiety Disorder 7 (GAD-7) | will be measured at baseline, 1 month, 3 months, and 6 months after enrollment (and start of intervention in the intervention arm)
  anxiety symptom measure; scores range from 0-21; higher scores are worse

CONTACTS AND LOCATIONS:
Overall Officials: Kari A Stephens, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington Primary Care, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made upon request after evaluation for appropriateness by principal investigator as an appropriate research request by individuals seeking to do further research. All data will be de-identified to protect participant privacy.
Supporting Information: Study Protocol, SAP
Time Frame: Sharing will occur after the publication of the final outcomes of the study are published and will be available for up to 7 years post completion of data collection.
Access Criteria: The requestor must provide acceptable research justification and appropriate permissions from their institutional to use the data requested for specific and detailed research purposes.

REFERENCES:
- [Background] Stephens, K. A., Ma, K., Keiser, B., Prado, M., Zhang, Y., West, I., Hsu, C., Anastas, T., Zbikowski, S., Waters, D., & Masterson, J. (2024, August). Improving chronic pain through use of a digital behavioral health app. Abstract and poster presented at the American Psychological Association Annual Convention, Seattle, WA.